CLINICAL TRIAL: NCT02021968
Title: A Phase 1 Evaluation of the Protective Efficacy of a Single Dose of the Live Attenuated Tetravalent Dengue Vaccine TV003 to Protect Against Infection With Attenuated DENV-2, rDEN2∆30-7169
Brief Title: Evaluating the Safety and Effectiveness of a Dengue Virus Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 287
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TetraVax-DV-TV003 vaccine (Experimental): Participants in this arm will receive a single injection of the TetraVax-DV-TV003 vaccine on Day 0 (study entry). On Day 180, participants will receive a single injection of the attenuated rDEN2∆30-7169 virus.
  Interventions: Biological: TetraVax-DV-TV003; Biological: rDEN2∆30-7169
- Placebo (Placebo Comparator): Participants in this arm will receive a single injection of placebo on Day 0 (study entry). On Day 180, participants will receive a single injection of the attenuated rDEN2∆30-7169 virus.
  Interventions: Biological: rDEN2∆30-7169; Biological: Placebo

INTERVENTIONS:
Biological: TetraVax-DV-TV003 — TetraVax-DV-TV003 is a live attenuated recombinant tetravalent dengue virus vaccine, which will be administered as a 0.5 mL dose containing 10^3.0 plaque forming units (PFUs) each of DENV-1, DENV-2, DENV-3, and DENV-4. It will be delivered by subcutaneous injection in the deltoid region of the upper arm.
  Other Names: TV003
  Arms: TetraVax-DV-TV003 vaccine
Biological: rDEN2∆30-7169 — The challenge virus, rDEN2∆30-7169, is a live recombinant attenuated DENV-2 candidate vaccine virus and will be administered as a 0.5 mL dose containing 10^3 PFUs of rDEN2∆30-7169. It will be delivered by subcutaneous injection in the deltoid region of the upper arm.
Biological: Placebo — The placebo vaccine is the vaccine diluent 1X L-15, which will be administered as a 0.5 mL dose delivered by subcutaneous injection in the deltoid region of the upper arm.
  Arms: Placebo

SUMMARY:
Dengue viruses can cause dengue illness ranging from a mild illness to life-threatening disease. The purpose of this study is to evaluate the protective effectiveness of a dengue virus vaccine in healthy adults.

DETAILED DESCRIPTION:
There are 4 types of dengue virus (DENV-1, DENV-2, DENV-3, and DENV-4); each can cause dengue illness ranging from a mild illness to life-threatening disease. More than 2 billion persons in tropical and subtropical regions of the world are at risk for acquiring dengue, which is why development of a dengue vaccine is a top public health priority.

The purpose of this study is to evaluate the ability of a single dose of TetraVax-DV-TV003 (TV003) vaccine to protect against infection with rDEN2∆30, an attenuated candidate DENV-2 vaccine.

This study will enroll healthy adults with no history of previous infection with a flavivirus (any of a group of viruses that includes the dengue virus). Participants will be randomly assigned to receive either the TV003 vaccine or placebo vaccine on Day 0 (study entry). At Day 180, all participants will receive an injection of the "challenge" virus, rDEN2∆30, an attenuated (weakened) DENV-2 vaccine. For at least 30 minutes after each vaccination, participants will remain in the study clinic to be monitored for any adverse effects of the vaccines. Participants will record their temperature at least 3 times a day for 16 days after the first and second vaccinations.

In addition to vaccination visits at Day 0 and Day 180, participants will attend study visits at Day 2, 4, 6, 8, 10, 12, 14, 16, 21, 28, 56, 90, 150, 182, 184, 186, 188, 190, 192, 194, 196, 201, 208, 236, 270, and 360. At all study visits, participants will give a medical history and undergo a blood collection; at most study visits, participants will undergo a physical examination. Female participants will have a pregnancy test at select study visits.

ELIGIBILITY:
Inclusion Criteria:

* Good general health as determined by physical examination, laboratory screening, and review of medical history
* Available for the duration of the study, approximately 26 weeks after second inoculation
* Willingness to participate in the study as evidenced by signing the informed consent document
* Females Only: Female participants of childbearing potential willing to use effective contraception. Reliable methods of contraception include: hormonal birth control, condoms with spermicide, diaphragm with spermicide, surgical sterilization, intrauterine device, and abstinence (6 months or more since last sexual encounter). All female participants will be considered having child-bearing potential except for those with hysterectomy, tubal ligation, tubal coil (at least 3 months prior to vaccination), or post-menopausal status documented as at least 1 year since last menstrual period.

Exclusion Criteria:

* Females Only: Currently pregnant, as determined by positive beta-human choriogonadotropin (HCG) test, breast-feeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the requirements of the study protocol
* Screening laboratory values of Grade 1 or above for absolute neutrophil count (ANC), alanine aminotransferase (ALT), and serum creatinine as defined in the study protocol.
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant participating in the trial or would render the participant unable to comply with the protocol
* Any significant alcohol or drug abuse in the past 12 months which has caused medical, occupational, or family problems, as indicated by participant history
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the last 6 months)
* HIV infection, by screening and confirmatory assays
* Hepatitis C virus (HCV) infection, by screening and confirmatory assays
* Hepatitis B virus (HBV) infection, by hepatitis B surface antigen (HBsAg) screening
* Any known immunodeficiency syndrome
* Use of anticoagulant medications
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 28 days prior to or following vaccination. Immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg prednisone equivalent per day for 14 days or longer.
* Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 28 days following vaccination
* Asplenia
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 28 days following vaccination
* History or serologic evidence of previous dengue virus infection or other flavivirus infection (e.g., yellow fever virus, St. Louis encephalitis virus, West Nile virus)
* Previous receipt of a flavivirus vaccine (licensed or experimental)
* Anticipated receipt of any investigational agent in the 28 days before or after vaccination
* Participant has definite plans to travel to a dengue endemic area during the study
* Refusal to allow storage of specimens for future research

Inclusion Criteria for Second Vaccine

* Good general health as determined by physical examination and review of medical history
* Available for the duration of the study, approximately 26 weeks after the second dose
* Willingness to participate in the study as evidenced by signing the informed consent document
* Females Only: Female participants of childbearing potential willing to use effective contraception for the duration of the trial. Reliable methods of contraception include: hormonal birth control, condoms with spermicide, diaphragm with spermicide, surgical sterilization, intrauterine device, and abstinence (6 months or more since last sexual encounter). All female participants will be considered having child-bearing potential except for those with hysterectomy, tubal ligation, tubal coil (at least 3 months prior to vaccination), or post-menopausal status documented as at least 1 year since last menstrual period.

Exclusion Criteria for Second Vaccine

* Anaphylaxis or angioedema following the first dose of vaccine
* Females Only: Currently pregnant, as determined by positive beta-HCG test, breast-feeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the requirements of the study protocol
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant participating in the trial or would render the participant unable to comply with the protocol
* Any significant alcohol or drug abuse in the past 12 months which has caused medical, occupational, or family problems, as indicated by participant history
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the last 6 months)
* HIV infection, by screening and confirmatory assays
* HCV infection, by screening and confirmatory assays
* HBV infection, by HBsAg screening
* Any known immunodeficiency syndrome
* Use of anticoagulant medications
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 42 days prior to or following vaccination. Immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg prednisone equivalent per day for 14 days or longer.
* Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 28 days following vaccination
* Asplenia
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 28 days following vaccination
* Anticipated receipt of any other investigational agent in the 28 days before or after vaccination
* Participant has definite plans to travel to a dengue endemic area during the study
* Refusal to allow storage of specimens for future research

Other Treatments and Ongoing Exclusion Criteria

The following criteria will be reviewed on Study Days 28 and 56 following each vaccination. If any become applicable during the study, the participant will not be included in further immunogenicity evaluations, as of the exclusionary visit. The participant will, however, be encouraged to remain in the study for safety evaluations for the duration of the study.

* Use of any investigational drug or investigational vaccine other than the study vaccine during the 28-day period after vaccination
* Chronic administration (14 days or longer) of steroids (defined as prednisone equivalent of greater than or equal to 10 mg per day), immunosuppressants, or other immune-modifying drugs initiated during the 28-day period after vaccination (topical and nasal steroids are allowed)
* Receipt of a licensed vaccine during the 28-day period after vaccination
* Receipt of immunoglobulins and/or any blood products during the 28-day period after vaccination
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Protection against viremia induced by rDEN2∆30, determined by rDEN2∆20-7169 titer | Measured through Day 196
  Participants will receive rDEN2∆30-7169 at Day 180. Viremia caused by rDEN2∆30-7160 will be measured through Day 196. Blood samples will be obtained from all participants on Days 180, 182, 184, 186, 188, 190, 192, 194, and 196, and the titer of rDEN2∆20-7169 will be determined.
Frequency of TV003 and rDEN2∆30-7169-related adverse events (AEs), as classified by both severity and seriousness, through active and passive surveillance | Measured through participants' last study visit on Day 360
Dengue virus neutralizing antibody titer | Measured through participants' last study visit on Day 360
  Seropositivity to each serotype will be defined as a PRNT50 of greater than or equal to 1:10 by Day 90 (TV003) and by Day 270 (rDEN2∆30-7169).

OTHER OUTCOMES:
Frequency of viremia following TV003 vaccination | Measured through Day 16 visit
Quantity of viremia following TV003 vaccination | Measured through Day 16 visit
Duration of viremia following TV003 vaccination | Measured through Day 16 visit
Determine if peak neutralizing antibody (NAb) titer against DENV-2 following TV003 vaccination or NAb titer against DENV-2 measured at Day 180 correlates with protection against viremia, rash, and/or neutropenia following inoculation with rDEN2∆30-7169 | Measured through Day 208
  Neutralizing antibodies will be measured through Day 180 following vaccination with TV003; viremia, rash, and neutropenia elicited by DEN2∆30-7169 will be measured from Day 180 through Day 208

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research (CIR), Johns Hopkins School of Public Health; Beth Kirkpatrick, MD, Principal Investigator — University of Vermont
Locations (2):
- United States (2):
  - Center for Immunization Research (CIR), Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland
  - University of Vermont Vaccine Testing Center, Burlington, Vermont

REFERENCES:
- [Derived] Hanley JP, Tu HA, Dragon JA, Dickson DM, Rio-Guerra RD, Tighe SW, Eckstrom KM, Selig N, Scarpino SV, Whitehead SS, Durbin AP, Pierce KK, Kirkpatrick BD, Rizzo DM, Frietze S, Diehl SA. Immunotranscriptomic profiling the acute and clearance phases of a human challenge dengue virus serotype 2 infection model. Nat Commun. 2021 May 24;12(1):3054. doi: 10.1038/s41467-021-22930-6. PMID 34031380
- [Derived] Nivarthi UK, Swanstrom J, Delacruz MJ, Patel B, Durbin AP, Whitehead SS, Kirkpatrick BD, Pierce KK, Diehl SA, Katzelnick L, Baric RS, de Silva AM. A tetravalent live attenuated dengue virus vaccine stimulates balanced immunity to multiple serotypes in humans. Nat Commun. 2021 Feb 17;12(1):1102. doi: 10.1038/s41467-021-21384-0. PMID 33597521
- [Derived] Larsen CP, Whitehead SS, Durbin AP. Dengue human infection models to advance dengue vaccine development. Vaccine. 2015 Dec 10;33(50):7075-82. doi: 10.1016/j.vaccine.2015.09.052. Epub 2015 Sep 28. PMID 26424605